CLINICAL TRIAL: NCT00097292
Title: TrialNet Pathway to Prevention of T1D
Status: Recruiting | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: NHStudy (IND); UC4DK117009 (NIH); UC4DK106993 (NIH)
Record Dates: First submitted 2004-11-19; First posted 2004-11-22 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: "at risk" for developing type 1 diabetes; T1DM; T1D; juvenile diabetes; Type 1 Diabetes TrialNet; TrialNet
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Annual Re-Testing/Annual Metabolic Monitoring: Participants will be monitored annually for risk of type 1 diabetes.
- Semi-Annual Metabolic Monitoring: Participants will be monitored every six months for risk of type 1 diabetes

SUMMARY:
Rationale:

The accrual of data from the laboratory and from epidemiologic and prevention trials has improved the understanding of the etiology and pathogenesis of type 1 diabetes mellitus (T1DM). Genetic and immunologic factors play a key role in the development of T1DM, and characterization of the early metabolic abnormalities in T1DM is steadily increasing. However, information regarding the natural history of T1DM remains incomplete. The TrialNet Natural History Study of the Development of T1DM (Pathway to Prevention Study) has been designed to clarify this picture, and in so doing, will contribute to the development and implementation of studies aimed at prevention of and early treatment in T1DM.

Purpose:

TrialNet is an international network dedicated to the study, prevention, and early treatment of type 1 diabetes. TrialNet sites are located throughout the United States, Canada, Finland, United Kingdom, Italy, Germany, Sweden, Australia, and New Zealand. TrialNet is dedicated to testing new approaches to the prevention of and early intervention for type 1 diabetes.

The goal of the TrialNet Natural History Study of the Development of Type 1 Diabetes is to enhance our understanding of the demographic, immunologic, and metabolic characteristics of individuals at risk for developing type 1 diabetes.

The Natural History Study will screen relatives of people with type 1 diabetes to identify those at risk for developing the disease. Relatives of people with type 1 diabetes have about a 5% percent chance of being positive for the antibodies associated with diabetes. TrialNet will identify adults and children at risk for developing diabetes by testing for the presence of these antibodies in the blood. A positive antibody test is an early indication that damage to insulin-secreting cells may have begun. If this test is positive, additional testing will be offered to determine the likelihood that a person may develop diabetes. Individuals with antibodies will be offered the opportunity for further testing to determine their risk of developing diabetes over the next 5 years and to receive close monitoring for the development of diabetes.

DETAILED DESCRIPTION:
Detailed Description:

The Pathway to Prevention Study is conducted in two parts:

* Screening
* Monitoring (annual and semi-annual depending on risk)

In Screening , a simple blood test is done to screen for the presence of diabetes-related biochemical autoantibodies (GAD and mIAA). Additional autoantibodies ICA, IA-2A, and ZnT8A will also measured in individuals positive for mIAA. ICA, IA-2A, and ZnT8A will be measured in individuals positive for GAD. Participants can go to a TrialNet Clinical Center, Affiliate, or request a screening kit to have their blood drawn by a local physician or laboratory. Participants will be provided with their screening results within 4-6 weeks.

If autoantibodies are present, participants will be invited to have additional testing to determine their average risk of developing diabetes over the next 5 years. Participants that are single autoantibody positive will be re-tested annually for the development of multiple autoantibodies. Multiple autoantibody positive participants will undergo an eligibility visit which will include an Oral Glucose Tolerance Test (OGTT), re-testing for biochemical and islet cell autoantibodies if needed, and measurement of HbA1c.

Multiple autoantibody positive individuals with a normal glucose tolerance and an HbA1c < 6.0% will be asked to come for follow-up on annual basis; multiple autoantibody positive individuals with an abnormal glucose tolerance or an HbA1c ≥ 6.0%will be asked to come for follow-up visits on semi-annual basis.

Participants will be monitored for possible progression towards type 1 diabetes and may be offered the opportunity to enter into a prevention study such (e.g., Oral Insulin prevention study) or an early treatment study if they are diagnosed with type 1 diabetes while participating in the Natural History Study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 2 to 45 years old who have an immediate family member with type 1 diabetes (such as a child, parent, or sibling)
* Individuals 2-20 years old who have an extended family member with type 1 diabetes (such as a cousin, niece, nephew, aunt, uncle, grandparent, or half-sibling)
* Those aged 2 years to 45 years who are not family members and are known to have 1 or more islet antibodies

Exclusion Criteria:

To be eligible a person must not:

* Have diabetes already
* Have previous or current use of medications for the control of hyperglycemia/diabetes.
* Currently be using immunosuppressive or immunomodulatory agents (topical and inhaled agents are acceptable)
* Have known severe active diseases, and/or diseases which are likely to limit life expectancy or lead to the use of chronic immunosuppressive or immunomodulatory therapies during the course of the study

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: First and second/third degree relatives of individuals with type 1 diabetes.
Sampling Method: Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2004-02-01 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Development of type 1 diabetes | Monitoring is provided once or twice annually depending on risk level
  The primary outcome is the development of diabetes as defined by the American Diabetes Association (ADA) based on glucose testing, or the presence of symptoms and unequivocal hyperglycemia.

SECONDARY OUTCOMES:
Metabolic and Autoantibody Assessments | Metabolic and Autoantibody assessments are provided once or twice annually depending on risk level
  Oral Glucose Tolerance Test (OGTT) HbA1c Autoantibodies: ICA, IA-2A, GAD65A, mIAA, ZnT8A

CONTACTS AND LOCATIONS:
Overall Officials: Kevan Herold, M.D., Study Chair — Yale University
Locations (22):
- United States (17):
  - Childrens Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Riley Hospital for Children, Indiana University, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Benaroya Research Institute, Seattle, Washington
- Walter and Eliza Hall Institute, Parkville, Victoria, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- University of Turku, Turku, Finland
- Vita-Salute San Raffaele University, Milan, Italy
- University of Bristol, Bristol, United Kingdom

REFERENCES:
- [Background] Diabetes Prevention Trial--Type 1 Diabetes Study Group. Effects of insulin in relatives of patients with type 1 diabetes mellitus. N Engl J Med. 2002 May 30;346(22):1685-91. doi: 10.1056/NEJMoa012350. PMID 12037147
- [Background] Gale EA, Bingley PJ, Emmett CL, Collier T; European Nicotinamide Diabetes Intervention Trial (ENDIT) Group. European Nicotinamide Diabetes Intervention Trial (ENDIT): a randomised controlled trial of intervention before the onset of type 1 diabetes. Lancet. 2004 Mar 20;363(9413):925-31. doi: 10.1016/S0140-6736(04)15786-3. PMID 15043959
- [Background] Atkinson MA, Eisenbarth GS. Type 1 diabetes: new perspectives on disease pathogenesis and treatment. Lancet. 2001 Jul 21;358(9277):221-9. doi: 10.1016/S0140-6736(01)05415-0. PMID 11476858
- [Background] Verge CF, Gianani R, Kawasaki E, Yu L, Pietropaolo M, Jackson RA, Chase HP, Eisenbarth GS. Prediction of type I diabetes in first-degree relatives using a combination of insulin, GAD, and ICA512bdc/IA-2 autoantibodies. Diabetes. 1996 Jul;45(7):926-33. doi: 10.2337/diab.45.7.926. PMID 8666144
- [Background] Bingley PJ, Christie MR, Bonifacio E, Bonfanti R, Shattock M, Fonte MT, Bottazzo GF, Gale EA. Combined analysis of autoantibodies improves prediction of IDDM in islet cell antibody-positive relatives. Diabetes. 1994 Nov;43(11):1304-10. doi: 10.2337/diab.43.11.1304. PMID 7926304
- [Derived] Martinenghi S, Merolla A, Grogan P, Bianconi E, Senni E, Goncharova A, Massara F, Ragogna F, Bazzigaluppi E, Pastore MR, Bonfanti R, Bosi E. Prevention of diabetic ketoacidosis in relatives screened for islet autoantibodies and followed up in the TrialNet Pathway to Prevention study at a single institution in Italy. Diabetologia. 2025 Sep;68(9):1889-1898. doi: 10.1007/s00125-025-06461-z. Epub 2025 May 29. PMID 40439773
- [Derived] Triolo TM, Pyle L, Broncucia H, Armstrong T, Yu L, Gottlieb PA, Steck AK. Association of High-Affinity Autoantibodies With Type 1 Diabetes High-Risk HLA Haplotypes. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1510-e1517. doi: 10.1210/clinem/dgab853. PMID 34850014
- [Derived] Evans-Molina C, Sims EK, DiMeglio LA, Ismail HM, Steck AK, Palmer JP, Krischer JP, Geyer S, Xu P, Sosenko JM; Type 1 Diabetes TrialNet Study Group. beta Cell dysfunction exists more than 5 years before type 1 diabetes diagnosis. JCI Insight. 2018 Aug 9;3(15):e120877. doi: 10.1172/jci.insight.120877. eCollection 2018 Aug 9. PMID 30089716
- [Derived] Ferrara CT, Geyer SM, Evans-Molina C, Libman IM, Becker DJ, Wentworth JM, Moran A, Gitelman SE, Redondo MJ; Type 1 Diabetes TrialNet Study Group. The Role of Age and Excess Body Mass Index in Progression to Type 1 Diabetes in At-Risk Adults. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4596-4603. doi: 10.1210/jc.2017-01490. PMID 29092051
- [Derived] Bosi E, Boulware DC, Becker DJ, Buckner JH, Geyer S, Gottlieb PA, Henderson C, Kinderman A, Sosenko JM, Steck AK, Bingley PJ; Type 1 Diabetes TrialNet Study Group. Impact of Age and Antibody Type on Progression From Single to Multiple Autoantibodies in Type 1 Diabetes Relatives. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2881-2886. doi: 10.1210/jc.2017-00569. PMID 28531305
- [Derived] Herold KC, Usmani-Brown S, Ghazi T, Lebastchi J, Beam CA, Bellin MD, Ledizet M, Sosenko JM, Krischer JP, Palmer JP; Type 1 Diabetes TrialNet Study Group. beta cell death and dysfunction during type 1 diabetes development in at-risk individuals. J Clin Invest. 2015 Mar 2;125(3):1163-73. doi: 10.1172/JCI78142. Epub 2015 Feb 2. PMID 25642774
- See also: TrialNet Study Group — http://www.diabetestrialnet.org
- See also: Type 1 Diabetes Clinical Trials — https://www.niddk.nih.gov/about-niddk/research-areas/diabetes/type-1-diabetes-special-statutory-funding-program/special-diabetes-program-clinical-trials-recruiting-patients-families
- See also: American Diabetes Association — http://www.diabetes.org
- See also: Juvenile Diabetes Research Foundation International — http://www.jdrf.org